CLINICAL TRIAL: NCT03995433
Title: EARLY-MYO-CMR-II (EARLY Assessment of MYOcardial Tissue Characteristics by CMR in NSTEMI) Registry
Brief Title: EARLY-MYO-CMR-II Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EARLY-MYO-CMR-II
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Non-ST-Segment Elevation Myocardial Infarction (NSTEMI)
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this registry is to depict the myocardial tissue characteristics in NSTEMI patients by CMR and other cardiac imaging modalities and to assess the prognostic value of imaging-derived indices. Information will be collected prospectively in about 2000 NSTEMI patients in 10 sites. Subjects will be followed for up to 5 years.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, observational registry study of NSTEMI patients that undergo CMR examination. Information of other cardiac imagings and clinical outcomes are also prospectively collected in the database. This project will establish a prospective registry of 2000 NSTEMI patients in 10 sites with follow-ups of up to 5 years.

The aim of the project will be as following:

1. To investigate myocardial pathological features and functional changes in NSTEMI patients.
2. To identify CMR-derived indices that are associated with adverse clinical outcomes.
3. To compare CMR with other alternative cardiac imaging modalities (i.e., echocardiography or SPECT) on prognostic prediction in NSTEMI patients.
4. To compare myocardial tissue characteristics and functional changes in STEMI (data derived from EARLY-MYO-CMR) and NSTEMI patients.
5. To verify GRACE Score classification in NSTEMI from CMR imaging view.

ELIGIBILITY:
Inclusion Criteria:

NSTEMI patients who have had CMR imaging performed and have provided written consent.

Patient older than 18 years old with non-ST-segment elevation myocardial infarction (NSTEMI):

1. Ischemic symptoms (chest pain or equivalent) at rest ≥ 10 minutes within 24 hours of randomization,
2. One of the two following criteria:

   1. New ST-segment depression ≥ 0.1 mV (≥1 mm), or transient (< 30 minutes) ST-segment elevation ≥ 0.1 mV (≥ 1 mm) in at least 2 contiguous leads on the electrocardiogram,
   2. Elevation of cardiac biomarkers within 24 hours of randomization, defined as elevated troponin T, troponin I, or CK-MB level above upper limit of normal,
3. Patients who have had CMR imaging performed and have agreed to comply with the follow up requirements.

Exclusion Criteria:

1. Patient who is unable to comply with the follow-up schedule.
2. Patient who has any medical conditions that in the opinion of the investigators will not be appropriate to participate in the study.
3. Patient has a life expectancy of less than 6 months due to any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSTEMI patients undergo CMR examination are eligible for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-05-08 (Actual); Primary Completion 2019-07-08 (Estimated); Study Completion 2019-12-09 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events(MACE) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University.
Locations (1):
- Ren Ji Hospital Affliated to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided